CLINICAL TRIAL: NCT07241390
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Event-Driven Study to Investigate the Effect of Orforglipron on the Incidence of Major Adverse Cardiovascular Events in Participants With Established Atherosclerotic Cardiovascular Disease and/or Chronic Kidney Disease
Brief Title: A Study of Orforglipron (LY3502970) on Cardiovascular Outcomes in Adults With Atherosclerotic Cardiovascular Disease and/or Chronic Kidney Disease (ATTAIN-Outcomes)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27771; J2A-MC-GZPW (Other: Eli Lilly and Company); 2025-523123-22-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Atherosclerosis Cardiovascular Disease; Chronic Kidney Disease
Keywords: Heart Disease; Kidney Disease; Outcomes; Stroke
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Diseases; Kidney Diseases; Stroke | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orforglipron (Experimental): Participants will receive orforglipron orally + standard of care
  Interventions: Drug: Orforglipron
- Placebo (Placebo Comparator): Participants will receive placebo orally + standard of care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970
  Arms: Orforglipron
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure cardiovascular outcomes with orforglipron compared with placebo in participants with atherosclerotic cardiovascular disease (ASCVD) and/or chronic kidney disease (CKD). Participation in the study will last about 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Have established ASCVD and/or CKD

Exclusion Criteria:

* Have type 1 diabetes
* Have had a major heart condition within 60 days prior to screening
* Have New York Heart Association Functional Classification Class IV heart failure

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7140 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2031-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of Composite Endpoint of Major Cardiovascular Events | Baseline up to end of study (about 5 years)
  Composite endpoint includes nonfatal myocardial infarction, nonfatal stroke, hospitalization or urgent visit due to heart failure, coronary revascularization, or all-cause death

SECONDARY OUTCOMES:
Time to First Occurrence of Composite Endpoint of Major Cardiovascular and Kidney Events | Baseline up to end of study (about 5 years)
  Composite endpoint includes nonfatal myocardial infarction, nonfatal stroke, hospitalization or urgent visit due to heart failure, coronary revascularization, ≥40% sustained decline in estimated glomerular filtration rate (eGFR), end-stage kidney disease, or all-cause death
Change from Baseline in Total eGFR Slope | Baseline up to end of study (about 5 years)
Time to Onset of Type 2 Diabetes | Baseline up to end of study (about 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (553):
- Argentina (59):
  - Instituto de Investigaciones Clínicas Bahia Blanca, Bahía Blanca
  - CONEXA Investigacion Clinica S.A., Buenos Aires
  - Buenos Aires Macula S.A, Buenos Aires
  - CIPREC, Buenos Aires
  - Instituto Médico Especializado (IME), Buenos Aires
  - Cicemo Srl, Buenos Aires
  - Cardiología Palermo, Buenos Aires
  - Nefra Mansilla, Buenos Aires
  - Consultorio Medico Investigador Principal Dr Besada, Buenos Aires
  - Glenny Corp. S.A., Buenos Aires
  - Organizacion Medica de Investigacion, Buenos Aires
  - Stat Research S.A., Buenos Aires
  - Investigaciones Medicas Imoba Srl, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires
  - CEMEDIC, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - CEMEDIAB, C.a.b.a.
  - CEDIC, CABA
  - Instituto de Cardiología "Juana F. Cabral", Corrientes
  - Centro Diabetológico Dr. Waitman, Córdoba
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - Centro Medico Privado San Vicente Diabetes, Córdoba
  - Instituto Médico DAMIC, Córdoba
  - Hospital Italiano de Córdoba, Córdoba
  - Sanatorio Esperanza, Esperanza
  - CIPADI - Centro Integral de Prevencion y Atencion en Diabetes, Godoy Cruz
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - Centro de Salud Renal Junín, Junín
  - CIMeL, Lanús
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata
  - Instituto de Cardiología Wolff, Mendoza
  - CER medical Institute, Quilmes
  - DIM Clínica Privada, Ramos Mejía
  - Instituto Médico Río Cuarto, Río Cuarto
  - Fundacion Estudios Clinicos, Rosario
  - Fundación Innovaciencia, Rosario
  - INECO Neurociencias Oroño, Rosario
  - Instituto Especialidades de la Salud Rosario, Rosario
  - Instituto Médico Catamarca IMEC, Rosario
  - Instituto Médico Fundación Grupo Colaborativo Rosario Investigación y Prevención Medica, Rosario
  - Instituto de Investigaciones Clinicas Rosario, Rosario
  - Laboratorio de Hemostasia y Trombosis, Rosario
  - Hospital Provincial del Centenario, Rosario
  - Clínica de Nefrología, Urología y Enfermedades Cardiovasculares, S3000epv
  - Santa Maria de la Salud Centro Medico, San Isidro
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman
  - Corporación Médica San Martín, San Martín
  - Centro Modelo de Cardiología, San Miguel de Tucumán
  - Investigaciones Clínicas Tucumán, San Miguel de Tucumán
  - Go Centro Medico San Nicolás, San Nicolás
  - Centro de Diagnóstico y Rehabilitación (CEDIR), Santa Fe
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
  - Centro de Salud e Investigaciones Médicas, Santa Rosa
  - Sanatorio San Martin, Venado Tuerto
  - Instituto de Investigaciones Clinicas Zarate, Zárate
- Australia (15):
  - Nightingale Research, Adelaide
  - Paratus Clinical Research Western Sydney, Blacktown
  - Box Hill Hospital, Box Hill
  - Royal Brisbane and Women's Hospital, Brisbane
  - Paratus Clinical Research Canberra, Bruce
  - Emeritus Research, Camberwell
  - Nightingale Research - Frankston, Frankston
  - Canberra Hospital, Garran
  - Barwon Health, Geelong
  - Life Clinical Research, Ipswich
  - Fusion Clinical Research, Norwood
  - USC Clinical Trials Sunshine Coast, Sippy Downs
  - USC Clinical Trials Brisbane (South Bank), South Brisbane
  - University of Sydney - Charles Perkins Centre, Sydney
  - Innovate Clinical Research, Waitara
- Austria (8):
  - VIVIT, Feldkirch
  - Medizinische Universität Graz, Graz
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Cardio Metabolic Centre, Mattersburg
  - Private Practice - Dr. Evelyn Fliesser-Gorzer, Sankt Stefan ob Stainz
  - Klinik Hietzing, Vienna
  - Herz Zentrum Währing - Innere Medizin und Kardiologie | Alle Kassen und Privat, Vienna
  - Klinik Floridsdorf, Vienna
- Belgium (15):
  - Imelda General Hospital, Bonheiden
  - Algemeen Ziekenhuis klina, Brasschaat
  - Cliniques universitaires Saint-Luc, Brussels
  - Ziekenhuis Oost-Limburg, Campus St.-Jan, Genk
  - Jessa Ziekenhuis, Hasselt
  - Jan Yperman Ziekenhuis, Ieper
  - Kormont, Kluisbergen
  - AZ Groeninge Campus Kennedylaan, Kortrijk
  - UZ Leuven, Leuven
  - Centre Hospitalier Régional de la Citadelle, Liège
  - CHU Tivoli, Louvière
  - AZ Sint-Maarten, Mechelen
  - Doc at Sea, Middelkerke
  - Az Damiaan vzw, Ostend
  - AZ Delta vzw, Roeselare
- Brazil (34):
  - Centro de Pesquisa Clinica do Coracao, Aracaju
  - Hospital Universitário João de Barros Barreto, Belém
  - NUPEC - Cardio, Belo Horizonte
  - University Center of Belo Horizonte - Campus Buritis, Belo Horizonte
  - AngioKormann Blumenau, Blumenau
  - Hospital Universitário São Francisco de Assis - Bragança Paulista, Bragança Paulista
  - Chronos Pesquisa Clínica, Brasília
  - Instituto de Pesquisa clinica de Campinas, Campinas
  - Centro de Pesquisa Sao Lucas, Campinas
  - Loema Instituto de Pesquisa Clinica, Campinas
  - Hospital Universitário Maria Aparecida Pedrossian, Campo Grande
  - Hospital Universitário, Canoas
  - Cline Research Center, Curitiba
  - Instituto de Ensino e Pesquisa Clinica do Ceara, Fortaleza
  - Private Practice - Dr.Miguel N. Hissa, Fortaleza
  - CECIP - Centro de Estudos do Interior Paulista, Jaú
  - Centro de Pesquisa Clínica de Marília - CPCLIM, Marília
  - CHN - Complexo Hospitalar de Niterói, Niterói
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - Hospital Ana Nery (HAN) - Salvador, Salvador
  - Obras Sociais Irma Dulce, Salvador
  - Centro Multidisciplinar de Estudos Clinicos, São Bernardo do Campo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - Centro Internacional de Pesquisa Clínica (CIPES), São José dos Campos
  - CPHosp Medicina, Ensino e Pesquisa (CPQuali), São Paulo
  - CPCLIN, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - Hospital das Clinicas FMUSP, São Paulo
  - Instituto de Molestias Cardiovasculares de Tatui, Tatuí
  - CEDOES, Vitória
  - Integral Pesquisa e Ensino, Votuporanga
- Bulgaria (9):
  - Medical Center New Polyclinic Gabrovo, Gabrovo
  - Medical Center Tonus 2013, Pazardzhik
  - UMBAL "Kaspela", Plovdiv
  - University Multiprofile Hospital for Active Treatment "Pulmed", Plovdiv
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi" EAD, Plovdiv
  - MC Rusemed, Rousse
  - "University Multiprofile Hospital for Active Treatment "Aleksandrovska"" EAD", Sofia
  - Diagnostic Consultative Center Aleksandrovska, Sofia
  - Medical Center Berbatov, Yambol
- Canada (19):
  - Centricity Research Brampton Endocrinology, Brampton
  - Cambridge Cardiac Care Centre, Cambridge
  - Ecogene-21, Chicoutimi
  - Premier Clinical Trial Network, Hamilton
  - The Wharton Medical Clinic Clinical Trials Inc, Hamilton
  - THEO Medical Concorde, Laval
  - G A Research Associates, Moncton
  - Applied Medical Informatics Research, Montreal
  - CHU de Quebec - Université Laval - Hotel Dieu de Quebec, Québec
  - Diex Recherche Quebec, Québec
  - C.I.C. Joliette, Saint-Charles-Borromée
  - Bluewater Clinical Research Group Inc., Sarnia
  - Heart Health Institute - Scarborough Office, Scarborough
  - Kidney Care Centre - Surrey, Surrey
  - Diex Recherche Inc. Division Trois-Rivieres, Trois-Rivières
  - Clinical Research Solutions - Kitchener, Waterloo
  - Winchester District Memorial Hospital, Winchester
  - Glanz Medicine Professional Corporation, Windsor
  - Seven Oaks General Hospital, Winnipeg
- China (25):
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Pinggu District Hospital, Beijing
  - China-Japan Union Hospital, Changchun
  - Changde First People's Hospital, Changde
  - Changzhou Second People's Hospital, Changzhou
  - Sichuan Provincial People's Hospital, Chengdu
  - 2nd Affiliated Hospital Chongqing Medical University, Chongqing
  - Guangdong Provincial People's Hospital, Guangzhou
  - Zhujiang Hospital, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The First Hospital of Harbin Medical University, Harbin
  - Jinan Central Hospital, Jinan
  - Jingjiang People's Hospital, Jingjiang
  - Jingzhou Central Hospital, Jingzhou
  - Lishui Central Hospital, Lishui
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi
  - Zhongshan Hospital,Fudan University, Shanghai
  - Jiading District Central Hospital, Shanghai
  - The Second Affiliated Hospital Of Shantou University Medical College, Shantou
  - Renmin Hospital of Wuhan University, Wuhan
  - Shaanxi provincial people's hospital, Xi'an
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - Zigong First People's Hospital, Zigong
- Colombia (11):
  - Fundacion Cardiomet Cequin, Armenia
  - Clinica de la Costa S.A.S., Barranquilla
  - Corazon IPS, Barranquilla
  - IPS Centro Científico Asistencial S.A.S, Barranquilla
  - Hospital Universitario Mayor Méderi, Bogotá
  - Bluecare Salud S.A.S, Bogotá D.C.
  - IPS Centro Médico Julián Coronel S.A.S, Cali
  - Fundación Oftalmológica de Santander FOSCAL, Floridablanca
  - IPS Médicos Internistas de Caldas, Manizales
  - Fundación Centro Médico COMETA, Pasto
  - Fundación Centro De Investigaciones Clinicas Ips Cardiomet Pereira, Pereira
- Czechia (14):
  - Diacentrum Brandys n.L. s.r.o., Brandýs nad Labem
  - Kardio Chlumec, Chlumec nad Cidlinou
  - KardioInt s.r.o., České Budějovice
  - MUDr. Alena Vachova, České Budějovice
  - DIKa Centrum, Havířov
  - Kardiologie KarMa, Jablonec nad Nisou
  - MUDr. Sabina Palova, Jílové u Prahy
  - MUDr. Tomas Edelsberger, Krnov
  - MUDr. Miroslav Koliba s.r.o., Ostrava
  - MUDr. Jana Parkanyiova, Prague
  - Milan Kvapil s.r.o., Diabetologicka ambulance, Prague
  - Praglandia s.r.o, Prague
  - Centrum Kardiovaskularni Mediciny, Prague
  - Diabetologie a endokrinologie, J.Venerová, Prague
- Estonia (4):
  - Private Practice - Dr. Liina Viitas, Pärnu
  - Center for Clinical and Basic Research AS, Tallinn
  - Estendo Private Clinic, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
- France (13):
  - Centre Hospitalier Universitaire - Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Bois-Guillaume
  - Chu Gabriel Montpied, Clermont-Ferrand
  - Chu Grenoble Alpes, La Tronche
  - Centre Hospitalier Louis Pasteur, Le Coudray
  - Hôpital Edouard Herriot, Lyon
  - Groupe Hospitalier de la Région de Mulhouse et Sud Alsace - Hôpital Emile Muller, Mulhouse
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes, Nantes
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur, Nice
  - Pitie Salpetriere University Hospital, Paris
  - CHU Rangueil, Toulouse
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Bretonneau, Tours
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (8):
  - Zentrum fur klinische Forschung - Köln, Cologne
  - Die Bocholder Hausärzte, Essen
  - Klinisches Forschungszentrum Dr. Hagemann am Hausarztzentrum am Germaniaplatz, Essen
  - Medizentrum Essen Borbeck, Essen
  - medicoKIT, Goch
  - Diabeteszentrum Hamburg West, Hamburg
  - RED-Institut GmbH, Oldenburg
  - Studienzentrum Brinkum - Torsten Drescher & Dr. Lars Pohlmeier, Stuhr
- Greece (8):
  - Athens Medical Center - Psychikon branch, Athens
  - Alexandra General Hospital of Athens, Athens
  - Athens Medical Center, Athens
  - University Hospital of Ioannina, Ioannina
  - Iatriko Paleou Falirou Medical Center, Palaió Fáliro
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki
  - European Interbalkan Medical Center, Thessaloniki
- Hungary (15):
  - DRC Gyógyszervizsgáló Központ, Balatonfüred
  - Szent Margit Rendelintézet, Budapest
  - ClinDiab Kft., Budapest
  - PVN Kutató Kft, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Cardiogeneral Egészségügyi Kft., Budapest
  - Újpesti Egészségközpont, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - CRU Hungary Kft., Encs
  - KomplexLabor Kecskemét, Kecskemét
  - Kistarcsai Flor Ferenc Korhaz, Kistarcsa
  - Szabolcs Szatmár Bereg Vármegyei Oktatókórház, Nyíregyháza
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
  - Regia Med Kft, Székesfehérvár
  - Zala Megyei Szent Rafael Kórház, Zalaegerszeg
- India (20):
  - Gujarat Endocrin Pvt Ltd, Ahmedabad
  - Life Care Hospital and Research Centre, Bangalore
  - KLES Dr. Prabhakar Kore Hospital & M.R.C, Belagavi
  - Belagavi Institute of Medical Sciences - Belagavi, Belagavi
  - All India Institute of Medical Sciences, Bhubaneswar
  - Endolife Speciality Hospitals, Guntur
  - Karnataka Medical College and Research Institute, Hubballi, Hubli
  - Osmania General Hospital, Hyderabad
  - K care Hospital, Kanpur
  - Nil Ratan Sircar Medical College and Hospital, Kolkata
  - Government Medical College - Kozhikode, Kozhikode
  - King George's Medical University, Lucknow
  - Central India Cardiology and Research Institute, Nagpur
  - Lata Mangeshkar Hospital - Digdoh, Nagpur
  - All India Institute of Medical Sciences (AIIMS) - Nagpur, Nagpur
  - G.B. Pant Institute of Postgraduate Medical Education & Research, New Delhi
  - National Heart Institute Delhi, New Delhi
  - All India Institute of Medical Sciences - Patna - Aurangabad Road, Patna
  - SMC Heart Institute and IVF Research Centre, Raipur
  - Rhythm Heart Institute - A Unit of SLPL, Vadodara
- Israel (16):
  - Assuta Ashdod Medical Center, Ashdod
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Hadassah Mount Scopus Medical Centre, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - ZIV Medical Center, Safed
  - Clalit Health Services - Sakhnin Community Clinic, Sakhnin
  - Diabetes Medical Center, Tel Aviv
  - Maccabi Healthcare Services, Tel Aviv
  - Yitzhak Shamir Medical Center, Ẕerifin
- Italy (14):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Asst Spedali Civili Di Brescia, Brescia
  - Azienda Ospedaliero Universitaria S.Anna, Ferrara
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Martino, Genova
  - Centro Cardiologico Monzino, Milan
  - Ospedale San Raffaele, Milan
  - Policlinico di Monza, Monza
  - A.O.U. Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Hospital Santa Maria della Misericordia in Perugia, Perugia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - IRCCS Policlinico San Donato, San Donato Milanese
- Japan (10):
  - Tokyo-Eki Center-building Clinic, Chūōku
  - NewHeart Watanabe Institute, Hamadayama, Suginami-ku
  - Rinku General Medical Center, Izumisano
  - Kobe City Medical Center General Hospital, Kobe
  - Yamanashi Prefectural Central Hospital, Kofu
  - Jinnouchi Hospital, Kumamoto
  - Yotsuya Internal Medicine Clinic, Shinjuku-ku
  - Higashi Takarazuka Satoh Hospital, Takarazuka
  - Uji-Tokushukai Medical Center, Uji
  - Japanese Red Cross Society - Wakayama Medical Center, Wakayama
- Lithuania (7):
  - Viešoji Istaiga Alytaus Poliklinika, Alytus
  - Kristavita, Jonava
  - UAB Hormodernus, Kaunas
  - Klinikiniai sprendimai, UAB, Kaunas
  - JSC Saules seimos medicinos centras, Kaunas
  - Kardiolitos Klinikos - Vilnius, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Malaysia (4):
  - Hospital Raja Permaisuri Bainun Ipoh, Ipoh
  - Hospital Raja Perempuan Zainab II, Kota Bharu
  - University Malaya Medical Centre, Lembah Pantai
  - Hospital Tuanku Jaafar Seremban, Seremban
- Mexico (36):
  - Centro de Atencion al Diabetico Actopan, Actopan
  - Medical Center Metas, Chihuahua City
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, S.C., Ciudad Madero
  - Instituto de Diabetes, Obesidad y Nutricion, Cuernavaca
  - Centro Para El Desarrollo de La Medicina Y de Asistencia Medica Especializada S.C., Culiacán
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Lahoja. Asociacion Para La Investigacion Y La Farmacovigilancia, Durango
  - Diseno y Planeacion en Investigacion Medica, Guadalajara
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad, Guadalajara
  - Unidad de Investigación Clínica y Atención Médica HEPA S.C., Guadalajara
  - Hermosillo Heart Team - Sinacor Hermosillo, Hermosillo
  - Investigación Médica Sonora, S.C., Hermosillo
  - Instituto Cardiovascular de León S.C., León
  - Centro de Investigacion en Artritis y Osteoporosis SC, Mexicali
  - RM Pharma Specialists - Unidad Especializada en Datos, Mexico City
  - Grupo Medico Camino Sc, Mexico City
  - Centro de Investigación Clinica Chapultepec, Mexico City
  - Gastrobariátrica Santa Fe, Mexico City
  - Hospital de Jésus, I.A.P., Mexico City
  - Centro Médico Nacional Siglo XXI, Mexico City
  - Hospital Juarez de Mexico, Mexico City
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Centro de Desarrollo Biomedico, Mérida
  - Medical Care and Research SA de CV, Mérida
  - Instituto Nacional de Cardiologia Ignacio Chavez, México
  - Centro de investigación y control metabólico, México
  - CEINV Salud, Monterrey
  - Cardiolink Clin Trials, Monterrey
  - Servicios de Oncología Medica Integral - Monterrey - José Benitez, Monterrey
  - UBAM Unidad Biomedica Avanzada Monterrey, Monterrey
  - Clínica García Flores SC, Monterrey
  - Centro de Investigacion Cardiovascular y Metabólica, Tijuana
  - FAICIC S. de R.L. de C.V., Veracruz
  - Integradora Multidisciplinaria Del Grijalva - Sinacor Villahermosa, Villahermosa
- Netherlands (22):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - EB Medical Research, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - OLVG Oost, Amsterdam
  - Amsterdam UMC, locatie AMC, Amsterdam
  - Gelre Ziekenhuis, Apeldoorn
  - Ziekenhuis Rijnstate, Arnhem
  - Het Van Weel-Bethesda Ziekenhuis - Ziekenhuis Dirksland, Dirksland
  - Slingeland Ziekenhuis, Doetinchem
  - Albert Schweitzer Ziekenhuis, locatie Dordwijk, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - Medische Centrum Leeuwarden, Leeuwarden
  - Alrijne Ziekenhuis, locatie Leiderdorp, Leiderdorp
  - Radboudumc, Nijmegen
  - Bravis Ziekenhuis, locatie Roosendaal, Roosendaal
  - Franciscus Gasthuis & Vlietland, Locatie Gasthuis, Rotterdam
  - Diakonessenhuis, locatie Utrecht, Utrecht
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Maxima Medisch Centrum, locatie Veldhoven, Veldhoven
  - VieCuri Medisch Centrum, locatie Venlo, Venlo
- New Zealand (6):
  - Aotearoa Clinical Trials, Auckland
  - Christchurch Heart Institute, Christchurch
  - Pacific Clinical Research Network - Waikato (PCRN Waikato), Hamilton
  - Pacific Clinical Research Network - Rotorua, Rotorua
  - Pacific Clinical Research Network - Wellington (PCRN Wellington), Upper Hutt
  - Aotearoa Clinical Trials - Whangarei, Whangarei
- Philippines (5):
  - Perpetual Succour Hospital, Cebu City
  - CARE CT Group, Dasmariñas
  - Health Cube Medical Clinics, Mandaluyong
  - Manila Doctors Hospital, Manila
  - Lorma Medical Center, San Fernando City
- Poland (20):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Zdrowie Osteo-Medic, Bialystok
  - Specderm Poznanska sp.j., Bialystok
  - IN VIVO, Bydgoszcz
  - Centrum Medyczne NEUROMED, Bydgoszcz
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Ambulatorium Sp. z o.o., Elblag
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - Clinical Best Solutions, Lublin
  - Centrum Medyczne "Diabetika", Radom
  - NZOZ Przychodnia Specjalistyczna Andrzej Wittek, Henryk Rudzki, Ruda Śląska
  - Poradnia AKA-MED Centrum Sp. z o.o., Ruda Śląska
  - Velocity Skierniewice Sp. z o.o., Skierniewice
  - Centrum Szybkiej Diagnostyki Kardiologicznej "Kardiomed" M. Żabówka E. Żabówka, Tarnów
  - Medon Clinical Research Sp. z o.o., Warsaw
  - Międzyleski Szpital Specjalistyczny w Warszawie, Warsaw
  - 4 Wojskowy Szpital Kliniczny z Polikliniką SPZOZ, Wroclaw
  - Samodzielny Publiczny Zespol Opieki Zdrowotnej w Wyszkow, Wyszków
  - Kardio Life, Włocławek
- Romania (20):
  - CMI Cardiologie - Dr. Mercea Corina Delia, Baia Mare
  - CMI DNBM Dr. Pop Lavinia, Baia Mare
  - Spitalul Clinic De Urgenta Prof Dr Agrippa Ionescu, Baloteşti
  - C.M.D.T.A. Neomed, Brasov
  - Nicodiab, Bucharest
  - Geea Medical Easy Diet, Bucharest
  - Centrul Medical NutriLife, Bucharest
  - Lotus-Med Tunari, Bucharest
  - CRN - Clinical Research Network, Bucharest
  - Diabet Med, Bucharest
  - Cardiomed Iași, Iași
  - Diabdana, Oradea
  - Dianutrilife Medica, Ploieşti
  - Clinica Korall, Satu Mare
  - Policlinica Astra Sibiu, Sibiu
  - SC Dentosim Queen SRL - Centrul Medical Diamed, Târgu Mureş
  - Mediab S.R.L., Târgu Mureş
  - Private Practice - Dr. Cristian Podoleanu, Târgu Mureş
  - Cabinet Medical Dr.Geru, Timișoara
  - Centrul Medical Medicalis, Timișoara
- Serbia (6):
  - Clinical Center of Serbia, Belgrade
  - General Hospital Krusevac, Kruševac
  - Institut Niška Banja, Niška Banja
  - General Hospital Sveti Luka, Smederevo
  - Sremska Mitrovica Health Centre, Sremska Mitrovica
  - Health Center Zajecar, Zaječar
- Slovakia (11):
  - Diacrin s.r.o., Bratislava
  - Medispektrum s.r.o, Bratislava
  - B. Braun Avitum - Galanta, Galanta
  - INTERN, s. r. o., Ilava
  - B.Braun Avitum - Pezinok, Pezinok
  - DENTAVIA, Poprad
  - DIA-MED CENTRUM s.r.o., Púchov
  - SPAOLO, s. r. o., Stará Turá
  - MUDr. Žáková, s.r.o. Vseobecna ambulancia pre dospelych, Trenčín
  - B. Braun Avitum - Dialyzacne stredisko Trstena, Trstená
  - MEDIVASA, Žilina
- South Africa (5):
  - TREAD Research, Cape Town
  - Soweto Clinical Trials Centre, Johannesburg
  - Paarl Research Centre, Paarl
  - Mediclinic Vergelegen, Sommerset West
  - Clinical Projects Research, Worcester
- South Korea (17):
  - The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si
  - Dong-A University Hospital, Busan
  - Pusan National University Yangsan Hospital, Busan
  - Daegu Catholic University Medical Center, Daegu
  - Hanyang University Guri Hospital, Guri-si
  - Chosun University Hospital, Gwangju
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Namdong-gu
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (16):
  - Centro Periférico de Especialidades Bola Azul, Almería
  - Hospital Universitario de La Ribera, Alzira
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario HM Monteprincipe, Boadilla del Monte
  - Hospital Ribera Polusa, Lugo
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitari Son Espases, Palma
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Quiron Infanta Luisa, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital de Alta Resolución de Utrera, Utrera
  - Hospital Clinico de Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Taiwan (15):
  - Changhua Christian Hospital, Changhua County
  - Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - Far Eastern Memorial Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
  - National Yang Ming Chiao Tung University Hospital, Yilan
- Thailand (3):
  - Faculty of Medicine Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Songklanagarind hospital, Hat Yai
- Tunisia (2):
  - Hopital Regional Mohamed Tahar Al Maamouri, Nabeul
  - Hopital Habib Thameur, Tunis
- Turkey (Türkiye) (14):
  - Adana Sehir Egitim ve Arastirma Hastanesi, Adana
  - Afyon Kocatepe Üniversitesi Tıp Fakültesi, Afyonkarahisar
  - Ankara Etlik City Hospital, Ankara
  - Akdeniz Universitesi Hastanesi, Antalya
  - Çanakkale Onsekiz Mart Üniversitesi, Çanakkale
  - Hitit Universitesi Corum Erol Olcok Egitim Ve Arastirma Hastanesi, Çorum
  - Eskisehir Osmangazi University, Eskişehir
  - Mehmet Akif Ersoy Research and Training Hospital, Istanbul
  - Erciyes Universitesi Tıp Fakultesi Hastaneleri, Kayseri
  - Kocaeli Üniversitesi, Kocaeli
  - Istanbul Kanuni Sultan Suleyman Egitim ve Arastirma Hastanesi, Küçükçekmece
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi, Malatya
  - Necmettin Erbakan University Meram Medical Faculty, Meram
  - Sakarya Training and Research Hospital, Sakarya
- Ukraine (19):
  - Regional Communal Non-commercial enterprise "Chernivtsi regional clinical hospital", Chernivtsi
  - Bazismed, Chernivtsi
  - Clinical Diagnostic Center, Ivano-Frankivsk
  - Institute of Endocrinology and Metabolism named after Komissarenko, Kiev
  - Kyiv City Endocrinological Center, Kyiv
  - Oleksandrivska City Clinical Hospital, Kyiv
  - Edelweiss Medics, Kyiv
  - Medical Center Ok!Clinic+, Kyiv
  - Medbud Clinic, Kyiv
  - ARTEM, Kyiv
  - Medical Center of Limited Liability Company "Medical Center "Consilium Medical", Kyiv
  - Center of Family Medicine Plus, Kyiv
  - Lviv City Clinical Hospital #4, Lviv
  - Branch "Center of Endocrinological Health" of "Lviv Regional Clinical Diagnostic Center", Lviv
  - PE "Poltava Regional Clinical Hospital n.a.M.V.Sklifosovsky PRC", Poltava
  - Zakarpattia Endoclinic, Uzhhorod
  - Medical Center Salutem, Vinnytsia
  - Vinnytsia Regional Clinical Endocrinology Dispensary, Vinnytsia
  - Communal Enterprise "Hospital #1" of Zhytomyr City Council, Zhytomyr
- United Kingdom (8):
  - FutureMeds - Birmingham, Birmingham
  - Layton Medical Centre, Blackpool
  - FutureMeds - Liverpool, Bromborough
  - Futuremeds-Newcastle, Newcastle
  - Newquay Health Centre, Newquay
  - The Adam Practice, Poole
  - Clifton Medical Centre, Rotherham
  - Rame Group Practice, Torpoint

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Orforglipron (LY3502970) on Cardiovascular Outcomes in Adults With Atherosclerotic Cardiovascular Disease and/or Chronic Kidney Disease (ATTAIN-Outcomes) — https://trials.lilly.com/en-US/trial/667755